CLINICAL TRIAL: NCT06430996
Title: Effects of Caffeinated Chewing Gum on 400-meter Performance and Fatigue Index of Sprinters: a Crossover Trial
Brief Title: Caffeinated Chewing Gum on 400-meter Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Hui Chiu (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113-2
Record Dates: First submitted 2024-04-08; First posted 2024-05-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Caffeine; Placebo
Keywords: exercise performance; fatigue index; α amylase
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): The participants chewing caffeine gum 10 minutes before exercise
  Interventions: Dietary Supplement: caffeine
- placebo gum (Placebo Comparator): The participants chewing placebo gum 10 minutes before exercise
  Interventions: Dietary Supplement: caffeine

INTERVENTIONS:
Dietary Supplement: caffeine — The participants chewing either caffeine Gum (CAF trial, containing 3 mg/kg of caffeine) or Placebo Gum (PL) for 10 minutes. After rested for 15 minutes, the participants underwent tests.
  Other Names: plocabo gum

SUMMARY:
20 trained sprinter were divided into caffeine Gum trial (CAF) and Placebo trial (PL) with a randomized, double-blind study design. The participants chewing either caffeine Gum (CAF trial, containing 3 mg/kg of caffeine) or Placebo Gum (PL) for 10 minutes. The outcomes are Running-Based Anaerobic Sprint Test and 400-meter sprint test was performed.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effect of caffeinated chewing gum on 400-meter sprint performance. 20 trained sprinter were divided into caffeine Gum trial (CAF) and Placebo trial (PL) with a randomized, double-blind study design. The participants chewing either caffeine Gum (CAF trial, containing 3 mg/kg of caffeine) or Placebo Gum (PL) for 10 minutes. After rested for 15 minutes, the participants underwent a Running-Based Anaerobic Sprint Test. After a 30-minute break, a 400-meter sprint test was performed. The blood lactate concentration were collected before and after 400-meter sprint from finger. Saliva samples were predicted to be collected before chewing gum, before the RAST, and after a 400-meter sprint. Saliva samples will be analyzed for caffeine and α-amylase concentrations in saliva.

ELIGIBILITY:
Inclusion Criteria:

* 6 years of professional short sprinting training
* 6 months of ongoing training, and
* 3 months of recovery from sports injuries such as strains and sprains.

Exclusion Criteria:

* Non-specialized sprinters.
* has not trained regularly for the past 6 months.
* has recovered from an athletic injury.
* less than 3 months of recovery from a sports injury, or participants with epilepsy, hypertension, hyperlipidemia, heart disease, arthritis, osteoporosis, brain injury, or a history of caffeine allergy.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Running-Based Anaerobic Sprint Test (RAST) | 15 minutes after intervention
  Measure the fatigue index (%)
400-meter sprinting | 30 minutes after RAST
  Measure the 400-meter completion time (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: ChihHui Chiu, PhD, Principal Investigator — Sport Science Research Center
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Only participant number and relevant experimental data are provided.

DOCUMENTS (1):
  • Study Protocol (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT06430996/Prot_000.pdf